CLINICAL TRIAL: NCT04964453
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 474121 in Healthy Japanese Male Subjects (Doubleblind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Men to Test How BI 474121 is Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1411-0012
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Healthy subjects were given a single dose of placebo tablet(s) matched to the active treatment, subjects receiving placebo were equally distributed across dose groups. Tablet(s) were taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: Placebo
- 2.5 mg BI 474121 (Experimental): Healthy subjects were given a single dose of 2.5 milligram (mg) of BI 474121 as a single (2.5 mg) uncoated tablet taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 474121
- 5 mg BI 474121 (Experimental): Healthy subjects were given a single dose of 5 milligram (mg) of BI 474121 as two (2.5 mg) uncoated tablets taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 474121
- 10 mg BI 474121 (Experimental): Healthy subjects were given a single dose of 10 milligram (mg) of BI 474121 as a single (10 mg) uncoated tablet taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 474121
- 20 mg BI 474121 (Experimental): Healthy subjects were given a single dose of 20 milligram (mg) of BI 474121 as two (10 mg) uncoated tablets taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 474121

INTERVENTIONS:
Drug: Placebo — Healthy subjects were given a single dose of placebo tablet(s) matched to the active treatment, subjects receiving placebo were equally distributed across dose groups. Tablet(s) were taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Arms: Placebo
Drug: BI 474121 — Healthy subjects were given a single dose of BI 474121 as a uncoated tablet(s) taken orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Arms: 10 mg BI 474121; 2.5 mg BI 474121; 20 mg BI 474121; 5 mg BI 474121

SUMMARY:
Safety, tolerability, and pharmacokinetics of BI 474121 will be assessed in healthy Japanese male using single rising oral doses in order to provide the basis for an ongoing clinical development of BI 474121 for the treatment of cognitive impairment in patients with Alzheimer's Disease and schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)) including body temperature, 12-lead electrocardiogram (ECG), and clinical laboratory tests at screening visit
* Japanese ethnicity, according to the following criteria:

  * born in Japan, have lived outside of Japan <10 years,
  * have parents and grandparents who are Japanese
  * Age of 20 to 45 years (inclusive) at screening visit
* Body mass index (BMI) of 18.5 to 25.0 kilogram per square meter (kg/m2) (inclusive) at screening visit
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication

  * Use of adequate contraception by any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration.
  * Vasectomized (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator at screening visit
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 millimetre of mercury (mmHg), or pulse rate outside the range of 50 to 90 beats per minute (bpm) at screening visit
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening visit
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator

  * Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
  * Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
  * Chronic or relevant acute infections including viral hepatitis, human immunodeficiency virus (HIV) and/or syphilis.
* History of cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a trial with a randomised within dose groups, placebo-controlled, double-blind, parallel group design to investigate safety, tolerability, and pharmacokinetics following single rising doses of BI 474121.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who were randomised and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (8.6) | 36.0 (8.4) | 27.0 (5.8) | 32.3 (9.0) | 36.5 (9.4) | 31.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 6 | 6 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 6 | 6 | 6 | 6 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events (AEs)
Description: Percentage of subjects with investigator-defined drug-related adverse events (AEs).
Time Frame: From the time of first administration of study medication until 168 hours (7 days) after time of administration, up to 8 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Percentage of participants | 25 | 0 | 16.7 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72 and 96 hours following drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were randomised and treated with at least one dose of study drug and who provided at least one pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/liter
Arm/Group | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanomole/liter | 289 (25.6) | 658 (21.2) | 1440 (15.4) | 2330 (25.4)

3. Secondary Outcome: Maximum Measured Concentration of BI 474121 in Plasma (Cmax)
Description: Maximum measured concentration of BI 474121 in plasma (Cmax).
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were randomised and treated with at least one dose of study drug and who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter
Arm/Group | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanomole/liter | 27.0 (20.6) | 54.3 (13.5) | 113 (11.2) | 193 (16.7)

ADVERSE EVENTS:
Time Frame: Adverse events: From the time of first administration of study medication until 168 hours (7 days) after time of administration, up to 8 days. All-cause mortality: From the time of first administration of study medication until end of trial, up to 15 days.
Description: Treated set (TS): all subjects who were randomised and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received.
Arm/Group | Placebo | 2.5 mg BI 474121 | 5 mg BI 474121 | 10 mg BI 474121 | 20 mg BI 474121
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 1/6 | 1/6 | 2/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | 2.5 mg BI 474121 (N=6) | 5 mg BI 474121 (N=6) | 10 mg BI 474121 (N=6) | 20 mg BI 474121 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT04964453/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04964453/SAP_001.pdf